CLINICAL TRIAL: NCT04720950
Title: The Impact of Morning or Evening Exercise on Total Energy Intake and Food Preference in Non-Exercising Adults.
Brief Title: The Impact of Morning or Evening Exercise on Food Intake
Acronym: TIME-Ex-Ulster
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Ulster (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: FCBMS-20-061
Record Dates: First submitted 2021-01-12; First posted 2021-01-22 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Obesity
Keywords: Energy intake; Time of day; Exercise; Circadian rhythms; Food preferences
MeSH Terms: conditions — Obesity; Motor Activity; Food Preferences | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Randomised crossover trial
Who Masked: Participant
Masking Description: True purpose of the study is blinded to participants.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Morning exercise (Experimental): 1 hour of exercise completed between 0800-1000
  Interventions: Other: Exercise
- Evening exercise (Experimental): 1 hour of exercise completed between 1800-2000
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — 1 hour of exercise on a motorised treadmill at 70% maximal heart rate

SUMMARY:
The beneficial effects of regular exercise on both physical and mental health are widely known; it is a pivotal component in the treatment and prevention of many metabolic disorders, including obesity. Exercise facilitates weight management, not only by increasing energy expenditure but through its effect on appetite regulation and, therefore, energy intake.

Multiple factors influence the effect of exercise on appetite regulation including body fat , gender, intensity and duration of exercise and levels of habitual physical activity . However, recently interest has grown around the impact time-of-day of exercise may have on appetite regulation . Subjective feelings of hunger follow a strong diurnal pattern, with feelings of hunger peaking in the evening and appearing lowest in the morning . Evening energy intake has been associated with increased total energy intake and body mass index Evening exercise could potentially counteract or lessen the evening hunger sensations and therefore reduce evening and total energy intake. The aim of this study is to investigate any changes in total energy intake, distribution of energy intake, and food preference on the day of and 24 -hours after a bout of moderate-intensity exercise completed in the morning or evening in a group of physically inactive adults. A total sample of 12 physically inactive adults aged 18-60 will be recruited on to the study. The study will take the form of a two-armed randomised controlled crossover trial consisting of two 48-hr overnight stays in the Human Intervention Studies Unit (HISU) at Ulster University, Coleraine, Northern Ireland. The participant information sheet will focus on the effect of morning and evening exercise on ambulatory blood pressure and exercise-induced feeling states to prevent the participants' knowledge of the true purpose of the study from influencing their feeding behaviours. Ambulatory blood pressure will be monitored for at least 24 hours after the exercise session and participants will be asked to complete questionnaires of exercise induced feeling states immediately before and after each exercise session. Participants will be briefed on the true purpose of the study following the study completion. During the visits, participants will be asked to perform 1 hour of exercise at 70% of their maximal heart rate on a motorised treadmill between either 0800-1000 or 1800-2000 on the first full day of the study appointment. Food will be provided ad libitum for the duration of the study. All food intake will be noted and covertly weighed and directly observed through security cameras in the HISU dining room and lounge areas to measure food-related behaviours, such as grazing or bingeing. A 24 hour dietary recall will be conducted at the end of each study appointment to validate recall against observed intake.

ELIGIBILITY:
Inclusion Criteria:

* Does not exercise regularly (as determined by International Physical Activity Questionnaire (IPAQ) short form.
* Able to perform 1 hour of moderate-intensity exercise on a treadmill.

Exclusion Criteria:

* Pregnancy/ lactation.
* Have significant dysphagia, gastric outlet obstruction, or any other factor which prevents the consumption of a meal.
* Have a significant food allergy or dietary restriction.
* Have a systemic or gastrointestinal condition that may affect food intake or preference.
* Taking medication or supplements that affect energy intake or appetite.
* Taking medication that affects blood pressure or heart rate.
* Have an irregular sleep or shift work patterns.
* Travel across > one time zone in the last month.
* Fitted with pacemaker
* Smokes or uses vaping products

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-05-31 (Estimated); Study Completion 2021-05-31 (Estimated)

PRIMARY OUTCOMES:
Total energy intake | Over 48 hours
  Covertly weighed food intake (kJ/day)

SECONDARY OUTCOMES:
Distribution of energy intake across the day | Over 48 hours
  Covertly weighed food intake (kJ/eating epochs)
Percentage energy intake from macronutrients | Over 48 hours
  % energy intake from fat, total carbohydrates, sugar, protein and fibre
Basal metabolic rate | Over 8 minutes after waking
  By indirect calorimetry
Ambulatory blood pressure | Over 24 hours
  Measured using Spacelabs 90217 ambulatory monitors
Exercise induced feelings state. | Change over 1 hour (pre exercise to post exercise)
  Measured using The Exercise Induced Feeling Inventory (EFI)
Validation of 24 hour dietary recall against observed intake | Over 48 hours
  Direct comparison between observed and reported food intake (kJ, % energy contribution from macronutrients)

CONTACTS AND LOCATIONS:
Locations (1):
- Human Intervention Studies Unit, Coleraine, N.Ireland, United Kingdom

IPD SHARING:
Plan to Share IPD: No